CLINICAL TRIAL: NCT00266578
Title: Effect of Swallowed Fluticasone Propionate on Eosinophilic Esophagitis; A Prospective, Randomized, Placebo-Controlled Trial
Brief Title: A Study Comparing Swallowed Flovent and Placebo in Patients With Eosinophilic Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marc Rothenberg (Other)
Responsible Party: Sponsor-Investigator, Marc Rothenberg, MD, PhD, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02-9-9; FAAN
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Fluticasone Propionate — Flovent vs. placebo daily for 3 months

SUMMARY:
The purpose of this study is assessing the efficacy of swallowed Flovent® vs. placebo for the treatment of eosinophilic esophagitis (EE).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for study by parent or guardian. Assent will be obtained from all minors 11 years of age and older.
* Age older than or equal to 3 years and younger than or equal to 30 years
* Endoscopic findings consistent with EE (edema, furrowing, exudates, rings)
* Histological findings to include proliferation of basal layer and peak eosinophil density ≥24 per high power field (400x). This degree of tissue eosinophilia has been shown to correlate well with poor-responsiveness to acid suppression therapy, suggesting it is a primary eosinophilic disease and not secondary to GERD[11].
* Allergy evaluation including skin-prick testing with multiple food antigens to insure elimination diet is not indicated.
* If allergic to specific foods, option to be on a minimum 3 months of elimination diet without detectable resolution by repeat endoscopy with biopsies demonstrating no improvement to disease.
* Patients enrolled at CCHMC will be under the direct care of Dr. Putnam or any of the other staff gastroenterologists at this institution who will supervise endoscopic procedures. Patients may also be enrolled at institutions other than CCHMC, but the diagnosis of EE must be validated by an expert pathologist in EE at CCHMC (Margaret Collins, MD).
* 20 additional patients without EE will be enrolled as unaffected controls for purposes of comparison with patients with EE. Enrollment pool will comprise patients undergoing routine upper endoscopy and having no identifiable pathology.

Exclusion Criteria:

* Patients with history of poor tolerance to FP, patients unable to cooperate with use of MDI, pregnant females, patients inhaling any corticosteroid for asthma, and patients with concurrent or recent (within 3 months) use of systemic steroids.

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2002-10; Primary Completion 2006-11 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Histologic remission | 5 years
  Histologic remission,defined by a peak eosinophil count of less than/equal to 1 eosinophil in all 400 fields in both the proximal and distal esophagus.

SECONDARY OUTCOMES:
Furrowing, Epithelial hyperplasia, clinical symptoms | 5 years
  Secondary outcome measures included presence of endoscopic furrowing, presence of epithelial hyperplasia, and presence of clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Marc E. Rothenberg, M.D., Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States